CLINICAL TRIAL: NCT05959083
Title: A Prospective, Multi-center, Post-marketing, Observational Study to Evaluate the Safety and Effectiveness of Upadacitinib in Chinese Adolescent and Adult Patients With Moderate to Severe Atopic Dermatitis (AD)
Brief Title: Real World Study of Oral Upadacitinib Tablets to Assess Adverse Events and Change in Disease Activity in Adolescent and Adult Chinese Participants With Atopic Dermatitis
Status: Active, not recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P21-702
Record Dates: First submitted 2023-07-17; First posted 2023-07-25 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Atopic Dermatitis (AD)
Keywords: Atopic Dermatitis (AD); Upadacitinib; RINVOQ
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Upadacitinib: Adolescent and adult participants will receive upadacitinib as prescribed by their physician irrespective of the study participation.

SUMMARY:
Atopic dermatitis (AD) is a skin condition that may cause a rash and itching due to inflammation of the skin. This study will assess how safe and effective upadacitinib is in treating AD in adolescent and adult Chinese participants.

Upadacitinib is an approved drug for treating AD. Approximately 200 adolescent and adult participants who are prescribed upadacitinib by their physician in accordance with local label will be enrolled in China.

Participants will receive upadacitinib as prescribed by their physician according to their routine clinical practice and local label. Participants will be followed up for approximately 24 months per participant and 30 days after last treatment dose for safety data collection.

There is expected to be no additional burden for participants in this trial. Participants will attend regular visits during the study at a hospital or clinic according to their routine clinical practice

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate to severe atopic dermatitis (AD) at the time of enrollment.
* Chinese adolescents (≥12 to <18 years of age with body weight of ≥40 kg) or adults (≥18 years of age) at the time of enrollment.
* Participants eligible for initiation of Upadacitinib treatment for AD, including any required screening tests indicated per China Label.
* The decision to prescribe Upadacitinib is made prior to and independently of study participation.

Exclusion Criteria:

* Participants who cannot be treated with Upadacitinib as per China label or by judgement of treating physician.
* Currently participating in any interventional research studies.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adolescent and adult Chinese participants with atopic dermatitis (AD) who are prescribed Upadacitinib by their physician according to their local label.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-08-18 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Incidence of Serious Infections | Up to approximately 25 months
  Incidence rate of serious infections in AD participants treated with Upadacitinib will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (18):
- China (18):
  - Peking University Third Hospital /ID# 257722, Beijing, Beijing Municipality
  - The First Affiliated Hospital Of Fujian Medical University /ID# 257725, Fuzhou, Fujian
  - Dermatology Hospital of Southern Medical University /ID# 261862, Guangzhou, Guangdong
  - The Eighth Affiliated Hospital, Sun Yat-sen universtiy /ID# 257737, Shenzhen, Guangdong
  - People's Hospital of Henan Province /ID# 257736, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technol /ID# 257724, Wuhan, Hubei
  - The First Hospital of China Medical University /ID# 257641, Shenyang, Liaoning
  - Second Affiliated Hospital of Xian Jiaotong University /ID# 257733, Xi'an, Shaanxi
  - Shandong Dermatological Hospital /ID# 257727, Jinan, Shandong
  - Huashan Hospital, Fudan University /ID# 256456, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine /ID# 257726, Shanghai, Shanghai Municipality
  - Shanghai Skin Disease Hospital /ID# 257719, Shanghai, Shanghai Municipality
  - Chengdu Second Municipal People's Hospital /ID# 257732, Chengdu, Sichuan
  - West China Hospital, Sichuan University /ID# 257720, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital /ID# 263898, Chengdu, Sichuan
  - Hangzhou First People's Hospital /ID# 261867, Hangzhou, Zhejiang
  - The second affiliated hospital of Zhejiang University school of medicine /ID# 257723, Hangzhou, Zhejiang
  - Ningbo First Hospital /ID# 263884, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=P21-702